CLINICAL TRIAL: NCT04353453
Title: A Prospective, Single-Center, Controlled Study to Evaluate the Performance of CardiacSense PPG Sensor in the CardiacSense1 Device
Brief Title: Study to Evaluate the Performance of CardiacSense PPG Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CardiacSense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL00201
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation
Keywords: Cardiology
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Study Procedure for Participants That Were Not in the Driving Group — Subjects were fitted with One lead Holter monitor and the CardiacSense1 watch simultaneously and were tested in the following condition:
  1. Sitting down for 10 minutes, walking for one minute and repeat this sequence twice at Indoor 28 ±3 degree Celsius.
  2. Sitting down for 10 minutes, walking for one minute and repeat this sequence twice at Indoor 22 ±3 degree Celsius.
  3. Sitting down for 10 minutes,outdoor walking for one minute and repeat this sequence four times At the end the devices were removed from the subject by the medical staff.The recorded data was downloaded for analysis by the Sponsor
Device: Study Procedure for Participants That Were Included in the Driving Group — Subjects were fitted with One lead Holter monitor and the CardiacSense1 watch simultaneously and were tested in the following condition:
  1. Sitting down for 10 minutes, walking for one minute and repeat this sequence twice at Indoor 28 ±3 degree Celsius.
  2. Sitting down for 10 minutes, walking for one minute and repeat this sequence twice at Indoor 22 ±3 degree Celsius.
  3. Going from the indoor facility to the car and driving for 30 minutes at least. Subject drove the car in city streets under light traffic conditions. At the end the devices were removed from the subject by the medical staff.The recorded data was downloaded for analysis by the Sponsor

SUMMARY:
study to evaluate the performance of the CardiacSense1's embedded PPG under different environmental and physical conditions

DETAILED DESCRIPTION:
The clinical study is a Prospective, Open, Single-Center, and Controlled Study to Evaluate the Performance of a PPG sensor in the CardiacSense1 device.

The CardiacSense1 is a wrist worn device designed to detect atrial fibrillation (AF). The AF detection of the device is based on a portable photoplethysmograph (PPG) sensor that is designed for continuous heart rate monitoring. The photoplethysmograph is a noninvasive circulatory signal related to the pulsatile volume of blood in the tissue.

Twenty (20) subjects (female and male) that do not suffer from atrial defibrillation and additional four (4) patients who are diagnosed as suffering from atrial fibrillation will be enrolled to the study.

Comparison of CardiacSense1 PPG individual peak detection to the corresponding recorded activity of an FDA-cleared ECG Holter, on a beat-by-beat basis will be performed on the following conditions:

All subjects will be exposed to 45 minutes of indoor standard office fluorescent light and 45 minutes to outdoor sunlight during mid-day. In addition, Subjects will be asked to walk for 1 minute once every 10 minutes and will be exposed to an indoor environment of 22±3 - 28±3 degree Celsius for 45 minutes and outdoor temperature of at least 15 degree Celsius, on the other 45 minutes.

4 Subjects will be tested in the following conditions: driving a car for 30 minutes; High wrist hair density subjects; Two subjects 65 y/o or older, two subjects 30 y/o or younger; Two subjects with BMI below 18.5 (underweight) and two subjects with BMI over 30 (Obesity); Two subjects with skin type 6 (Fitzpatrick) and two subjects with skin type 5; Four subjects with diagnosed persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Age of eighteen to eighty-five (18-85) years
* Ability and willing to sign informed consent form
* For subjects in groups other than Heart Arrhythmias- Self-declared not to be diagnosed with any arrhythmia
* Compliance with hair, age, BMI skin and heart arrhythmia variables as defined above

Exclusion Criteria:

* Concurrent enrollment in another device or drug trial that has not completed the primary endpoint or clinically interferes with the current study endpoints.
* Subject with low perfusion indicated by the watch
* Pregnant or breastfeeding woman (women of child-bearing potential must have a negative pregnancy test within screening period).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
PPG individual peak detection | 90 Minutes
  Comparison of CardiacSense1 PPG individual peak detection to the corresponding recorded activity of an FDA-cleared ECG Holter, on a beat-by-beat basis.
PPG and Holter ECG signals correlation | 90 Minutes
  Evaluation of the correlation between PPG signals and Holter ECG signals with respect to R-R signal intervals.

SECONDARY OUTCOMES:
signal intensity under different conditions | 90 minutes
  Examination of PPG signal optic parameters (LED current, LED intensity) and signal intensity under different conditions.
Adverse events | 90 minutes
  Rate of Adverse events related or unrelated to the study device.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
IPD is not available to other researchers